CLINICAL TRIAL: NCT06362980
Title: An Open-label, Single-arm, Investigator-initiated Phase I Clinical Study Evaluating BPI-1178 Capsules in Combination With Osimertinib Tablets in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer With EGFR Mutations
Brief Title: A Study With BPI-1178 and Osimertinib in Advanced Non-small Cell Lung Cancer Patients With EGFR Mutations
Acronym: EGFR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Center, China (Other)
Responsible Party: Principal Investigator, Puyuan Xing, Chief Medical Officer, National Cancer Center, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPI-1178-IIT01
Record Dates: First submitted 2024-03-28; First posted 2024-04-12 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: NSCLC
Keywords: NSCLC; EGFR Gene Mutation; BPI-1178; Osimertinib
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BPI-1178 plus Osimertinib treatment (Experimental): Patients will undergo treatment with a combination of BPI-1178 capsules and osimertinib tablets. Patients will orally receive a single dose of BPI-1178 (200 or 300 mg) capsules and osimertinib tablets (80 mg). After a 7-day washout period, continuous dosing will commence on the 8th day. During the continuous dosing phase, BPI-1178 capsules and osimertinib tablets will be administered once daily, with a treatment cycle consisting of 28 days.
  Interventions: Drug: BPI-1178; Drug: Osimertinib

INTERVENTIONS:
Drug: BPI-1178 — 200 or 300 mg, oral, QD
  Other Names: BPI-1178 capsule
Drug: Osimertinib — 80mg, oral, QD
  Other Names: Tagrisso

SUMMARY:
BPI-1178 is a novel, orally administered inhibitor of both cyclin-dependent kinase 4 (CDK4) and CDK6 kinase activity. This open-label investigator-initiated trial (IIT) phase I study was designed to evaluate the safety and efficacy of oral BPI-1178 in combination with osimertinib in patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) and epidermal growth factor receptor (EGFR) Mutations.

DETAILED DESCRIPTION:
This study is an open-label, single-arm, single-center clinical study initiated by the researcher. The plan is to enroll 20 patients with locally advanced or metastatic NSCLC harboring EGFR mutations. The study aims to assess the safety and conduct preliminary observations on the efficacy of BPI-1178 capsules in combination with osimertinib in treating locally advanced or metastatic EGFR mutation-positive NSCLC patients who have developed resistance to osimertinib.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible for this study:

1. Signed written informed consent and ability to comply with the scheduled visits and study procedures outlined in the protocol.
2. Age ≥ 18 years, any gender.
3. Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer (mainly adenocarcinoma) not suitable for curative surgery or radiation therapy.
4. ECOG Performance Status (ECOG PS) score of 0-1. Expected survival of at least 12 weeks.
5. Prior treatment with a third-generation EGFR tyrosine kinase inhibitor (TKI) targeted therapy, with radiological evidence of disease progression. The last treatment before enrollment must show radiological evidence of disease progression, intolerance to chemotherapy toxicity, or the patient being ineligible for standard treatment or unable to tolerate the current treatment regimen.
6. At least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria that has not been previously irradiated.
7. Tissue, plasma, or cytological samples collected after disease progression confirmed by imaging following treatment with a third-generation EGFR TKI, demonstrating an EGFR-positive gene mutation sensitive to EGFR TKI treatment (including exon 19 deletion, 21 L858R mutation, etc.), with or without T790M mutation.
8. Adequate organ and bone marrow function, with clinical laboratory test results meeting the following criteria:

   * Hematology: Neutrophils ≥ 1.5 × 10^9/L; Platelets ≥ 100 × 10^9/L; Hemoglobin (Hgb) ≥ 100 g/L;
   * Liver function: Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN) (≤3 × ULN for patients with Gilbert's syndrome); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × ULN;
   * Renal function: Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance rate (CCr, Cockcroft-Gault formula) ≥ 50 mL/min; Semi-quantitative urine testing (e.g., urine dipstick) result showing urine protein < 2+; patients with urine protein ≥ 2+ at baseline should undergo a 24-hour urine collection, and the protein content in the urine within 24 hours should be < 1g;
   * Coagulation function: Activated partial thromboplastin time (APTT) and international normalized ratio (INR) both ≤ 1.5 × ULN;
   * Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%;
   * At rest, male QTcF < 450 msec or female QTcF < 470 msec.
9. Ability to swallow oral medications.
10. Reproductive-age female patients must agree to use effective contraception throughout the study period until 60 days after discontinuing BPI-1178 and osimertinib. Female patients must have a negative pregnancy test result before the start of treatment or prove the absence of pregnancy possibility. Male patients must agree to use effective contraception throughout the study period until 120 days after discontinuing BPI-1178 and osimertinib.
11. Apart from stable Grade 2 peripheral neuropathy (CTCAE v5.0) and alopecia, any treatment-related clinical toxicity before enrollment must have recovered to baseline or Grade 1.
12. All patients must have sufficient mental capacity to understand the nature, significance of the study, and risks associated with the study.

Exclusion Criteria:

Subjects with any of the following cannot be included in this study:

1. History of prior or current use of anti-tumor drugs targeting CDK4/6.
2. Individuals with allergies or a history of severe allergic reactions.
3. Tissue, plasma, or cytological samples collected after radiological confirmation of disease progression, with testing confirming the presence of specific therapeutic targets such as anaplastic lymphoma kinase (ALK), BRAF V600E, or retinoblastoma (Rb) protein loss.
4. Received the last dose of anti-tumor treatment (chemotherapy, targeted therapy, investigational drugs, immunotherapy, tumor embolization, herbal medicine for anti-tumor purposes, etc.) within the 2 weeks preceding the start of study drug administration.
5. Presence of third-space effusion (such as significant pleural or abdominal fluid) that cannot be controlled by drainage or other methods.
6. Long-term use of steroids is required.
7. Unresolved hypokalemia and hypomagnesemia at the time of enrollment.
8. Meets any of the following criteria: Various clinically significant arrhythmias and conduction abnormalities, such as atrial fibrillation, complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 msec; various factors that may increase the risk of QT interval prolongation or arrhythmia events, such as symptomatic heart failure - New York Heart Association (NYHA) class II-IV, congenital long QT syndrome, Brugada syndrome, history of QT interval prolongation (male > 470 ms, female > 480 ms) or torsades de pointes (TdP), family history of long QT syndrome or unexplained sudden death before the age of 40, various concomitant medications that may prolong QT interval; within the 6 months before starting the study drug, had the following diseases, including unstable angina, myocardial infarction, cerebrovascular accident, pulmonary embolism, etc., or underwent cardiac revascularization surgery.
9. History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid treatment, or any clinically evident active interstitial lung disease.
10. Known active infections, such as hepatitis B (HBsAg positive and hepatitis B virus (HBV) DNA copy number ≥ 200 IU/ml), hepatitis C, and human immunodeficiency virus (HIV) infection.
11. Cannot be included if there has been a relapse or concurrent malignancy in the past 5 years. Cervical cancer treated with curative intent, non-melanoma skin cancer, superficial bladder tumors (non-invasive tumors), or cancer with no recurrence for 3 years after curative treatment can be considered for inclusion.
12. History of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
13. Various factors judged by the investigator to potentially affect the intake and absorption of BPI-1178 or osimertinib, including gastrointestinal factors (such as uncontrolled inflammatory gastrointestinal diseases, history of abdominal fistula or gastrointestinal perforation within 6 months, extensive small intestine resection requiring enteral or parenteral supplementation, inability to swallow, chronic diarrhea, intestinal obstruction, etc.).
14. Spinal cord compression, leptomeningeal metastases, or symptomatic brain metastases cannot be included. Asymptomatic patients with brain metastases may be allowed to participate under the following conditions: Asymptomatic brain metastases discovered during screening, determined by the investigator not to require steroids and/or local treatment; asymptomatic brain metastases treated with local therapy (such as radiation) with the patient discontinuing steroids and/or antiepileptic treatment for at least 7 days before the first administration of BPI-1178 in combination with osimertinib.
15. Major surgery (craniotomy, thoracotomy, or laparotomy) or severe unhealed wounds, ulcers, or fractures within the 4 weeks preceding the start of study drug administration.
16. Local radiation therapy for symptom relief within 1 week before the first administration of the study drug; bone marrow radiation therapy or extensive radiation therapy exceeding 30% within 4 weeks before the first administration of the study drug.
17. Presence of factors, according to the investigator's judgment, that may interfere with patient participation in the trial or the assessment of study results, such as substance abuse, alcohol addiction, medical, psychiatric illness, and social disorders, or any factors that the investigator deems the patient unsuitable for receiving the study drug (such as severe hypertension, diabetes, thyroid disease, severe infection, portal hypertension, cirrhosis, etc.). Patients who were unwilling or unable to comply with the requirements of this study protocol will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose-limiting toxicity (DLT) | From first dosing (Day 7) to Day 28 of Cycle 1 (28 days/cycle)
  DLT will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 15 months
  The ORR is defined as the proportion of subjects with the best overall response of complete response (CR) or partial response (PR).
Disease Control Rate (DCR) | Up to approximately 15 months
  DCR is defined as the proportion of subjects with the best overall response of complete response (CR), partial response (PR), or stable disease (SD).
Duration of Response (DoR) | Up to approximately 15 months
  In subjects with the best overall response of complete response (CR) or partial response (PR), it refers to the time from the initial occurrence of complete or partial response to the occurrence of disease progression or death for any reason (whichever comes first).
Progression-Free Survival (PFS) | Up to approximately 15 months
  PFS is defined as the duration from the first study treatment until the onset of disease progression or death from any cause for the subjects.
Overall Survival (OS) | Up to approximately 15 months
  OS is defined as the duration from the initial study treatment to death from any cause among the subjects.
Intracranial ORR (iORR) | Up to approximately 15 months
  The intracranial ORR is defined as the proportion of subjects with an intracranial best overall response of complete response (CR) or partial response (PR).
Intracranial DCR (iDCR) | Up to approximately 15 months
  The intracranial DCR is defined as the proportion of subjects with an intracranial best overall response of complete response (CR), partial response (PR), or stable disease (SD).
Intracranial DoR (iDoR) | Up to approximately 15 months
  In subjects with an intracranial best overall response of complete response (CR) or partial response (PR), it refers to the duration from the first initial occurrence of complete or partial response to the occurrence of intracranial disease progression or death for any reason (whichever comes first).
Intracranial Time to Progression (iTTP) | Up to approximately 15 months
  Intracranial TTP is defined as the duration from the initiation of the first study treatment to the occurrence of intracranial disease progression among the subjects.
Intracranial PFS (iPFS) | Up to approximately 15 months
  Intracranial PFS is defined as the duration from the first study treatment until the onset of intracranial disease progression or death from any cause for the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Puyuan Xing, Doctorate, Principal Investigator — Department of Medical Oncology, National Cancer Center, China
Locations (1):
- National Cancer Center, Beijing, China

IPD SHARING:
Plan to Share IPD: No